CLINICAL TRIAL: NCT05917184
Title: The Adapting Disease Specific Outcome Measures Pilot Trial for Telehealth in Myasthenia Gravis (ADAPT-teleMG)
Brief Title: The Adapting Disease Specific Outcome Measures Pilot Trial for Telehealth in Myasthenia Gravis
Acronym: ADAPT-teleMG
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Richard Nowak, Principal Investigator, Yale University
Other Study IDs: 2000030599; 1U54NS115054-01 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Myasthenia Gravis
Keywords: Neuromuscular; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Muscle weakness; Autoimmune Diseases; Immune System Diseases; Neuromuscular Junction Diseases; Outcome measures
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Muscle Weakness; Autoimmune Diseases; Immune System Diseases; Neuromuscular Junction Diseases | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurological Outpatients: Participants in this group will be recruited from the outpatient clinical population at participating MGNet sites. Treating physicians will make the initial determination of patients' potential eligibility to participate in the study.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — Two video telehealth visits will be conducted and recorded within 3 days of one another (+/- 1 day)

SUMMARY:
The goal of this pilot study is to determine the reliability of myasthenia gravis (MG) specific outcome measures obtained during virtual encounters with patients with myasthenia gravis. The main question it aims to answer is: Are MG-specific outcome measures obtained during virtual encounters reliable?

Participants will complete two virtual study visits in which they will be administered common MG-specific outcome measures and a newly developed outcome measure developed specifically for telemedicine assessments of MG patients.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the use of modified clinical assessments during telehealth visits for patients with Myasthenia Gravis (MG). The study will consist of 2 virtual telemedicine visits. A screening visit will be conducted to optimize the telemedicine environment, provide training on the telemedicine platform being used in the study, and collect demographic, medical history, and medication information. Participants who meet eligibility requirements will have a telemedicine visit (Visit 1) with a study doctor where assessments adapted for the telemedicine environment will be performed. Participants will also be asked to fill out questionnaires related to MG or their experience with telemedicine either online or with the study investigators. A second visit (Visit 2), conducted within 3 days (+/- 1 day), will replicate the assessments performed in V1. Visit 1 and Visit 2 will be recorded for later review by study team members. The investigators hope to establish the effectiveness of these clinical tools in order to better manage MG in the future in clinical care and research study visits.

ELIGIBILITY:
Inclusion Criteria:

* Has the capacity to understand and sign an informed consent form
* Diagnosed with acquired autoimmune MG based on clinical syndrome and seropositivity for MG associated autoantibodies (AChR binding, MuSK, or LRP4 antibodies), and/or a decremental response on repetitive nerve stimulation, positive single-fiber electromyography or positive edrophonium test
* Subject has been previously evaluated in a face-to-face clinical encounter at one of the participating study sites within the prior 3 years
* Primary language is English, or equivalent level of English language fluency
* Required disease severity range from asymptomatic-mild to moderate-severe as previously judged by the Investigator.

Exclusion Criteria:

* Inadequate technology for telehealth visits as assessed by the Investigator (e.g., no internet connection, no laptop/tablet with video capability, etc). Cellular phones are not acceptable. Subjects must use a laptop or tablet.
* Is unable or unwilling to comply with the study procedures, including video recording, or telehealth visit.
* Any significant medical/psychiatric condition that, in the opinion of the Investigator, may interfere with interpretation of subject evaluation(s) or protocol compliance
* Known pregnancy
* MGFA severity class IVb or V
* Concurrent participation in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 adult participants with a confirmed diagnosis of MG will be enrolled with a range of disease activity from approximately 7 MGNet clinical study sites
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Interrater reliability of the virtual Myasthenia Gravis Composite (MGC-v) score. | 3 days (+/- 1 day)
  Interrater reliability of the virtual Myasthenia Gravis Composite (MGC-v) score will be estimated between two independent rater assessments performed on Visit 1 (V1) and Visit 2 (V2). The MGC score is a validated, patient-reported 10-item assessment tool for evaluating the symptoms and signs of MG. Patient assessment includes self-report of impact (normal, mild, moderate, or severe) and is additionally weighted for clinical significance. Total score ranges from 0 to 50, with higher scores indicating a greater impact of MG on functional activities. A three point change is considered clinical meaningful. This brief assessment takes approximately 10 minutes to complete.
Intrarater reliability (test-retest reliability) of the MGC-v score. | 3 days (+/- 1 day)
  Interrater reliability of the virtual Myasthenia Gravis Composite (MGC-v) score will be estimated between two independent rater assessments performed on Visit 1 (V1) and Visit 2 (V2). The MGC score is a validated, patient-reported 10-item assessment tool for evaluating the symptoms and signs of MG. Patient assessment includes self-report of impact (normal, mild, moderate, or severe) and is additionally weighted for clinical significance. Total score ranges from 0 to 50, with higher scores indicating a greater impact of MG on functional activities. A three point change is considered clinical meaningful. This brief assessment takes approximately 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nowak, MD, MS, Principal Investigator — Yale University; Amanda Guidon, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No